CLINICAL TRIAL: NCT01656590
Title: High Protein Nutrition and Exercise Therapy (HPET) Plus Nocturnal Enteral Feeding (NEF) in Juvenile-onset Pompe Disease.
Brief Title: High Protein and Exercise Therapy Plus Nocturnal Enteral Feeding in Juvenile-onset Pompe Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAJ7305
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Glycogen Storage Disease Type II
Keywords: Pompe disease; Acid Maltase Deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High Protein and Exercise therapy along-with Nocturnal Enteral (Other)
  Interventions: Other: High Protein and Exercise Therapy along-with Nocturnal Enteral Feeding

INTERVENTIONS:
Other: High Protein and Exercise Therapy along-with Nocturnal Enteral Feeding — 1. High Protein and Moderate Carbohydrate Nutrition designed by our nutritionist for every patient based on his/her nutrition requirements, age & gender
  2. 500 cc Formula - Nutren Replete with Fiber overnight [8 hours] via gastrostomy tube
  3. Conditioning Exercise once daily

SUMMARY:
The research protocol will be submitted for approval to the institutional review board of Columbia University Medical Center. An attempt will be made to recruit at least 6 juvenile patients between the ages of 8 and 17, preferably who are still ambulatory.

Subjects meeting all eligibility criteria will undergo a full history and physical examination, including details of age of onset of symptoms, distribution and severity of muscle weakness, muscle function, pulmonary function, and nutritional status. Subjects will undergo an electrocardiogram (ECG), spirometry, muscule strength evaluation, exercise capacity, functional muscle tests, laboratory tests, and muscle biopsy. Quality of life will be assessed via SF 36 questionnaire. Functional ability and level of handicap will be assessed by Rotterdam handicap scale. Written informed consent will be obtained from all subjects.

All patients, who will have received enzyme replacement therapy (ERT) for at least 2 years, will be evaluated prior to institution of high protein nutrition and exercise therapy plus nocturnal enteral feeding (HPET + NEF)(baseline), then again at 3 months, 6 months and 12 months into treatment. The following parameters will be evaluated-

* Skeletal Muscle Function
* Biochemical parameters from collected blood sample Muscle Biopsy will be obtained at baseline and at 12 months. Biopsy specimens, obtained from thigh muscle at baseline and a repeat biopsy of the corresponding area of the other leg at 12 months, will be analyzed as follows:.
* Histology and electron microscopy
* Autophagic and lysosomal function evaluation
* Body composition Body mass index (BMI), body composition, lean body mass, and fat mass will be measured at each visit by bioelectric impedance analysis using BI-101Q RJL Systems, software 3.1b

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 8 to 17 years of age.
2. Diagnosis of Pompe disease; either by enzyme deficiency of muscle biopsy specimen or skin fibroblast culture, or homozygous or compound heterozygous for GAA mutation.
3. Muscle Function < grade 7 on Walton Scale.
4. Women of reproductive age (> 15 years) agree to use reliable methods of contraception during the study, if sexually active
5. Subject or legal representative is willing and able to provide written informed consent.

Exclusion Criteria:

1. Any intercurrent condition that may preclude accurate interpretation of study data
2. Obstructive pulmonary disease
3. Invasive ventilatory support
4. Noninvasive ventilatory support while awake and in an upright position
5. History of QTc prolongation > 450 msec for males and > 470 msec for females
6. Life expectancy < 1 year
7. History of allergy, sensitivity or any serious adverse reaction to rhGAA drug
8. Pregnancy
9. Current or recent drug or alcohol abuse.
10. Treatment with another investigational drug within 60 days of study start
11. Use of prohibited medication < 3 months prior to randomization
12. Otherwise unsuitable for the study in the opinion of investigator

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in muscle function | Baseline, 12 months
  Gross muscle function will be measured by the Walton Scale, the Timed Muscle Function Test and the Six-Minute Walk. Muscle strength will be measured by hand held dynamometer. Functional ability will be assessed by Rotterdam 9-item Handicap Scale.

SECONDARY OUTCOMES:
Change in pulmonary function (Vital capacity, forced expiration volume) | Baseline, 12 months
  The Pulmonary Function Test will be used to measure vital capacity (VC) and forced expiration volume (FEV1) to assess pulmonary function in sitting and supine positions.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred E Slonim, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States